CLINICAL TRIAL: NCT01346163
Title: A Phase1B Study: A Placebo Controlled Study of PF-03654746 Given as Add-On Treatment of Cognitive Deficits in Schizophrenia
Brief Title: Add On Treatment for Cognitive Deficits in Schizophrenia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Raquel E. Gur, M.D., Ph.D., University of Pennsylvania School of Medicine
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 809087
Record Dates: First submitted 2009-05-20; First posted 2011-05-02 (Estimated); Last update posted 2011-05-02 (Estimated); Status verified 2011-04

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Cognitive Impairment; Electrophysiology; H3 receptor antagonist
MeSH Terms: conditions — Schizophrenia; Cognitive Dysfunction | interventions — N-ethyl-3-fluoro-3-(3-fluoro-4-(pyrrolidinylmethyl)phenyl)cyclobutanecarboxamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PF-03654746 (Active Comparator): H3 receptor antagonist currently being developed for the treatment of cognitive impairment associated with schizophrenia (CIAS) as well as with Alzheimer's disease.
  Interventions: Drug: PF 03654746
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: PF 03654746 — All participants will receive 3 weeks of PF-03654746 and 3 weeks of placebo. PF-03654746 and placebo will be administered in a flexible titration regimen, beginning with 0.5 mg/d. If 0.5 mg/d is well tolerated, the dose will be increased to 1.0 mg/d after 5 days. If 1.0 mg/d is not well tolerated, the dose will be decreased to 0.5 mg/d, with the goal of achieving a stable dose of PF-03654746 within the first two weeks of dosing and avoiding further dose changes during the final week of dosing.
  Arms: PF-03654746
Other: Placebo — Placebo will be used as a comparator to the active arm.
  Arms: Placebo

SUMMARY:
This study will look at the impact of dosing as well as ongoing treatment with an investigation medication identified as PF-03654746, on cognitive and physiologic indicators of brain function. Data from this study will assist with the evaluation of the utility of functional magnetic resonance imaging, arterial spin labeling (ASL), and electrophysiologic measures in the detection of early signals of the effectiveness of medications developed to target cognitive impairment in schizophrenia. Safety and tolerability of PF-03654746 in this population will be also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

Initial Inclusion Criteria:

1. Subjects must be competent to provide informed consent to participate in a clinical trial before any trial-related procedures can take place;
2. Subjects must be willing and able to comply with scheduled visits, treatments, laboratory tests and other testing and study procedures;
3. Subjects who participate must be willing to remain in-patient for at least one week at the beginning of each treatment period and remain in the hospital until judged by the Investigator to be clinically stable and able to be discharged to outpatient status;
4. Subjects must be fluent in English and able to understand all study related materials;
5. Subjects must be between the ages of 18-40 (inclusive) and if Female be of non-childbearing potential;
6. Body Mass Index (BMI) 18 to 40 kg/m2 and a total body weight of at least 50 kg (110 lbs);

Psychiatric Inclusion Criteria:

1. Subjects must have a current DSM-IV-TR diagnosis of schizophrenia of Paranoid (295.30), Disorganized (295.10), Undifferentiated (295.90) or Residual Type (295.60);
2. Subjects must be receiving ongoing maintenance antipsychotic monotherapy with risperidone, olanzapine, quetiapine, ziprasidone, paliperidone or aripiprazole;
3. Subjects must be on a stable medication treatment regimen 2 months, including concomitant psychotropic medications;
4. Evidence of stable control of symptoms for 3 months (eg, no hospitalizations for schizophrenia, no increase in level of psychiatric care due to worsening of symptoms of schizophrenia);
5. No more than moderate severity rating (4) on any individual PANSS positive symptom item (P1, P3, P5, P6) or formal thought disorder (P2), with no more than two moderate items in total;
6. Calgary Depression Scale Score less than or equal to 10;
7. Subjects must have a minimal level of extrapyramidal symptoms as documented by a score on the ESRS-A Global Parkinsonism scale of 3;
8. Subjects must have an illness duration (from the time of diagnosis) of at least 1 year;
9. Subjects will meet the following cognitive performance criteria:

   1. Performance less than the maximum cutoff (in parentheses) for at least ONE of the following MCCB tests: (i.) Letter-number span (20); (ii.) Hopkins Verbal Learning Test (HVLT) total (31); and (iii.) Continuous Performance T- test (CPT) d-prime (3.47);
   2. Able to complete the Baseline MCCB validly as assessed by a certified MCCB test administrator;
   3. Standard score greater than or equal to 75 on the National Adult Reading Test (NART) or other IQ measure.

Exclusion Criteria:

1. Female subjects who still have child bearing potential and females who are breastfeeding;
2. History of febrile illness within 5 days prior to the first dose;
3. Any condition possibly affecting drug absorption (eg, gastrectomy);
4. Subjects who have a positive urine drug screen which cannot be explained by prescribed medications;
5. History of regular alcohol consumption exceeding 7 drinks/week for females or 14 drinks/week for men (1 drink = 5 ounces (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of hard liquor) within 6 months of screening;
6. Treatment with an investigational drug within 30 days or 5 half-lives preceding the first dose of study medication;
7. 12-lead ECG demonstrating QTc less than or equal to 450 msec at screening;
8. Subjects who are using disallowed concomitant medications and who will not be able to discontinue these concomitant medications prior to randomization;
9. Subjects who have taken hormone replacement therapy within 28 days or have taken an herbal remedy 7 days prior to the first dose of trial medication;
10. Subjects with other conditions that may increase the risk associated with trial participation or investigational product administration or may interfere with the interpretation of trial results, and in the judgment of the Investigator, would make the subject inappropriate for entry into this trial;
11. Subjects with serologic evidence of acute hepatitis or chronic hepatitis and subjects with known hepatitis C antibodies and elevated LFTs;
12. Subjects with AST and/or ALT 1.5xULN at the Screening Visit;
13. Subjects with a current DSM-IV axis I diagnosis other than schizophrenia;
14. Subjects with a concurrent psychiatric disorder other than schizophrenia coded on Axis I;
15. Subjects who have previously participated in a trial using PF-03654746;
16. Subjects who have DSM-IV defined psychoactive substance dependence (excluding nicotine dependence) within 12 months of screening or substance abuse within 3 months prior to Screening;
17. Subjects currently using illicit psychoactive substances as evidenced by positive urine toxicology screen (utox positive for cannabinoids will not be exclusionary due to the long elimination half life of these substances);
18. Subjects with evidence or history of mental retardation;
19. Subjects with significant risk of suicidal or violent behavior;
20. Subjects with a history of poor compliance;
21. Subjects who have received clozapine or monoamine oxidase inhibitors in the month prior to randomization;
22. Current treatment with haloperidol or other typical antipsychotic;
23. Current treatment (within 4 weeks) with psychotropic agents known to act at the GABA-A receptor, including benzodiazepines; sedative-hypnotics other than trazodone and chloral hydrate; carbamazepine, gabapentin, lamotrigine, and valproic acid;
24. Current treatment (within 4 weeks) with psychotropic agents known to effect cognition: amphetamine; barbiturates; lithium; MAOIs; methylphenidate;
25. Current treatment (within 4 weeks) with herbal preparations with possible psychotropic effects (eg, St. Johns wort, kava-kava, Valerian, S-Adenosyl Methionine [SAMe]);
26. Subjects with a history of seizures and or/seizure disorder, significant head injury/trauma, as defined by one or more of the following:

    1. Loss of consciousness (LOC) for more than 1 hour;
    2. Recurring seizures resulting from the head injury;
    3. Clear cognitive sequelae of the injury;
    4. Cognitive rehabilitation following the injury.
27. Subjects with a history of clinically significant neurological, metabolic, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, and/or urological disorders (eg, unstable angina, decompensated congestive heart failure, CNS infection or history of HIV seropositivity), which would pose a risk to the patient if they were to participate in the study or that might confound the results of the study. Active medical conditions that are minor or well controlled are not exclusionary if they do not affect risk to the patient or the study results. For example, the following are not exclusionary: a) stable and well controlled hypertension (BP normally 160/95 for at least 3 months); b) asthma (no serious attacks in the past year); c) hypothyroidism (T4 within normal limits for at least 1 year); and d) Type II diabetes (subjects with a reported HgbA1c outside of normal limits within the last 6 months should be reviewed with the study site Investigator);
28. Subject received ECT treatment within the last 6 months;
29. Prior participation in a clinical trial of any other psychotropic medication within 2 months;
30. Subjects with a history of treatment resistant schizophrenia;
31. Subjects with a history of Tardive dyskinesia (TD) or Neuroleptic Malignant Syndrome (NMS) as determined clinically by the Investigator;
32. Unwilling or unable to comply with the Lifestyle guidelines described in this Protocol;
33. Subjects with implanted metal;
34. Subjects with claustrophobia such that they are unable to tolerate MR scanning.
35. Subjects taking medication that inhibit CYP3A4 or CYP2D6

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2009-04; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
MATRICS Consensus Cognitive Battery | 13 - 15 Weeks

SECONDARY OUTCOMES:
ASL perfusion and performance on neurocognitive measures | 3 Weeks
fMRI activation parameters and performance on neurocognitive measures. | 3 weeks
ERP measures and performance on neurocognitive measures | 3 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Raquel P. Gur, M.D., Ph.D., Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: University of Pennsylvania Department of Neuropsychiatry Home Page — http://www.med.upenn.edu/bbl/